CLINICAL TRIAL: NCT05678985
Title: Choose to Move (Phase 4): Impact and Implementation Evaluation of a Program to Enhance Older Adult Physical Activity, Mobility and Health
Brief Title: Evaluating Impact and Implementation of Choose to Move (Phase 4)
Acronym: CTM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Active Aging Society (Other)
Responsible Party: Principal Investigator, Heather McKay, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H20-00780; PJT-169159 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2022-12-19; First posted 2023-01-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Aging; Mobility Limitation; Sedentary Behaviour; Loneliness; Social Isolation; Social Connectedness
Keywords: Older adults; Behaviour change; Physical inactivity; Mobility; Social connectedness; Loneliness; Effectiveness; Maintenance; Implementation; Adaptation; Acceptability; Feasibility; Fidelity; Dose
MeSH Terms: conditions — Mobility Limitation; Social Isolation; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Choose to Move (Experimental): CTM (Phase 4) is a 3-month, flexible, choice-based program for low active older adults that can be delivered in-person or online.
  CTM includes
  * One-on-One Consultation: Participants meet 1-on-1 with their activity coach at the start of the program to set goals and develop an action plan tailored to their abilities, interests and resources. Older adults can choose to participate in individual or group-based activities.
  * Group Meetings: Over the 3-months, participants will attend eight, 1-hour group-based meetings (up to 12 participants total) led by their activity coach. Meetings cover a discussion topic (health-related) and provide time and space for social connection between participants. Group meetings are held in person or online as public health restrictions and community preference dictate.
  Interventions: Behavioral: Choose to Move

INTERVENTIONS:
Behavioral: Choose to Move — As described under study arm description.

SUMMARY:
The objectives of this study are to: 1) evaluate whether Choose to Move (CTM) Phase 4 improves health outcomes in older adults who participate and 2) assess whether CTM Phase 4 is delivered as planned and what factors support or inhibit its delivery at scale.

CTM Phase 4 is a 3-month, choice-based program for low active older adults being scaled-up across British Columbia (BC), Canada. The goals of CTM are to enhance physical activity, mobility and social connectedness in older adults living in BC, Canada.

DETAILED DESCRIPTION:
Choose to Move (CTM) Phase 4 is a 3-month, choice-based program for low active older adults being scaled-up in phases across British Columbia (BC), Canada. Within CTM (Phase 4), trained activity coaches support older adults in two ways. First, in a one-on-one consultation, activity coaches help participants to set goals and create action plans for physical activity tailored to each person's interests and abilities. Older adults can choose to participate in individual or group-based activities. Second, activity coaches facilitate 8 group meetings with small groups of participants. Activity coaches and recreation departments across BC are trained and provided with resources to deliver CTM.

Objectives:

1. To assess the impact (effectiveness) of CTM (Phase 4) delivered at scale on the physical activity, mobility, and social connectedness of older adults (Part I - Impact Evaluation)
2. To assess whether CTM (Phase 4) was implemented as planned (fidelity) and investigate factors that support or inhibit its implementation at scale (Part II - Implementation Evaluation).

Study Design:

The investigators use a hybrid type 2 effectiveness-implementation (Curran et al 2012) pre-post study design to evaluate CTM. The investigators use multiple methods (quantitative and qualitative) and collect data at 0 (baseline), 3 (post-intervention), 6 (3 months post-intervention), 15 (12 months post-intervention) and 27 (24 months post-intervention) months to assess impact and implementation of CTM.

ELIGIBILITY:
Inclusion Criteria (older adults):

* ≥60 years of age
* demonstrate readiness for physical activity via the PAR-Q+ questionnaire, Get Active Questionnaire, or a letter of recommendation from their physician
* <150 min/week physical activity
* English speaking
* Able to connect to the Zoom or GoToMeeting platform via phone or internet in order to participate in virtual group meetings (for online programs only)

Exclusion Criteria (older adults):

* Previous participation in CTM

Inclusion Criteria (delivery partners):

* Activity coaches will be English speaking, British Columbia Recreation and Parks Association (BCRPA) registered older adult fitness leaders or kinesiologists who are delivering CTM at participating centres
* Recreation Managers and Coordinators affiliated with participating centres delivering CTM
* Provincial Partners (e.g., individuals/partners who make strategic and/or policy decisions) at partner organizations delivering Choose to Move

Activity Coach inclusion criteria:

* Able to connect to the Zoom or GoToMeeting platform via internet (video and audio required in order to see and hear participants) for online programs
* Able to connect to the Zoom or GoToMeeting platform via phone or internet in order to participate in virtual group meetings (for online programs only)
* Currently (or recently completed) participating in CTM evaluation

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | 0, 3, 6, 15, 27-months
  The single item physical activity questionnaire will be used to measure physical activity. Output variable is self-reported number of days/week ≥30 min physical activity in the past week (range 0-7).

SECONDARY OUTCOMES:
Change in capacity for mobility | 0, 3, 6, 15, 27-months
  Two items will assess participants' ability to walk a quarter of a mile and up 10 steps. The output variable is self-reported presence of mobility-disability (no/any difficulty walking 400m or climbing one flight of stairs).
Change in physical functioning | 0, 3, 6, 15, 27-months
  The Physical Functioning Subscale of the SF-36 will be used to assess the physical function aspect of mobility. The measure asks participants to rate if their health limits them in performing 10 different activities. The output variable is an average score (range 0-100) of physical functioning, where a higher score indicates a more favourable health state.
Change in mobility | 0, 3, 6, 15, 27-months
  The Mobility Assessment Tool-Short Form (MAT-sf) will be used to assess mobility. MAT-sf is a validated, short form video-animated tool to assess participant self-perception of mobility. Only participants with an internet connection are able to complete this measure. The output variable is a self-perception of mobility score (range 23.45-67.61) where a higher score indicates greater perceived mobility.
Change in loneliness | 0, 3, 6, 15, 27-months
  The three-item loneliness scale will be used to assess loneliness. Participants rate three aspects of loneliness. The output variable is loneliness score (range 3-9); lower scores indicate lower levels of loneliness.
Change in social isolation | 0, 3, 6, 15, 27-months
  A three-item questionnaire adapted from two questions on social contact frequency will be used to assess social isolation. The output variable is social isolation score (range 0-15); higher scores indicate lower levels of social isolation.
Change in social network | 0, 3, 6, 15, 27-months
  A six-item questionnaire will be used to assess social network. The output variable is an equally weighted sum (range 0-30) where higher scores indicate more social engagement.
Change in social connectedness | 0, 3, 6, 15, 27-months
  A single item will be used to assess sense of belonging as an indicator of social connectedness. The output variable is sense of belonging score (range 1-4) where lower scores indicate a stronger sense of belonging.
Change in sitting time | 0, 3, 6, 15, 27-months
  A five-item questionnaire will be used to assess change in sitting time (hours and minutes) each day in the following domains: (a) while travelling to and from places (e.g., work, shops); (b) while at work; (c) while watching television; (d) while using a computer at home; and (e) at leisure not including watching television (e.g., visiting friends, movies, eating out) on a weekday and a weekend day. The output variables are sitting hours per day across 5 domains.
Change in screen time | 0, 3, 6, 15, 27-months
  A single item will be used to assess screen time. The output variable is hours of screen time per day.
Change in health-related quality of life (EQ-5D-5L Profile) | 0, 3, 6, 15, 27-months
  Health status will be assessed using the EQ-5D-5L. Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. Responses are used to create a 5-digit number which will be used descriptively (11111 indicates no problems on any of the five dimensions whereas 55555 indicates extreme problems on all five dimensions).
Change in health-related quality of life (EQ-5D-5L Level Sum Score) | 0, 3, 6, 15, 27-months
  Health status (EQ-5D-5L Level Sum Score) will be assessed with the EQ-5D-5L. Participants report on mobility, self-care, usual activities, pain/discomfort and anxiety/depression on a scale from 1-5 (level of perceived problems) for each item. The Level Sum Score uses the 5-digit profile to create a numeric score, with scores ranging from 5-25 (lower levels indicate lower levels of perceived problems).
Change in health-related quality of life (EQ-5D-5L Visual Analogue Scale) | 0, 3, 6, 15, 27-months
  Health status will be assessed with the EQ-5D-5L visual analogue scale. Participants report on their health on a visual analogue scale from 0 (worst health) to 100 (best health).

OTHER OUTCOMES:
Reach-individual | 3-months
  The number of participants engaged in the intervention will be obtained from program records.
Reach-organizational | 3-months
  The number of organizations and activity coaches delivering the intervention will be obtained from program records.
Dose delivered | 3-months
  The amount of intervention delivered will be assessed via survey (designed in house). Lower scores indicate that a lower dose of the intervention was delivered than planned.
Fidelity (survey) | 3-months
  Fidelity to planned delivery will be assessed via survey (designed in house). Higher scores indicate better adherence to planned delivery.
Fidelity (interview/focus group) | 3-months
  Fidelity to planned delivery will be assessed via interview/focus group.
Participant responsiveness (survey) | 3-months
  Program satisfaction will be assessed via participant survey (designed in house). Higher scores indicate higher participant satisfaction with the intervention.
Participant responsiveness (interview) | 3-months
  Program satisfaction will be assessed via interview.
Adaptation (survey) | 3-months
  Adaptation of the intervention and its delivery will be assessed via survey (designed in house).
Adaptation (interview/focus group) | 3-months
  Adaptation of the intervention and its delivery will be assessed via interview/focus groups.
Contextual factors influencing implementation (survey) | 3-months
  Contextual factors influencing implementation (community level factors, provider characteristics, characteristics of the innovation, the prevention delivery system, organizational capacity and the prevention support system) will be assessed via survey (designed in house).
Contextual factors influencing implementation (interview/focus group) | 3-months
  Contextual factors influencing implementation (community level factors, provider characteristics, characteristics of the innovation, the prevention delivery system, organizational capacity and the prevention support system) will be assessed via interviews/focus groups.
Cost | 3-months
  Program delivery costs will be recorded using a cost capture template.
Change in Organizational Readiness (Organizational Readiness Rubric) | 0, 3-months
  Organizational readiness (OR) will be assessed via survey (Organizational Readiness Rubric; ORR). The ORR comprises 14 items, each scored from 1-5. Higher mean scores indicate greater organizational readiness.
Change in Organizational Readiness (Readiness for Organizational Change Scale) | 0, 3-months
  Organizational readiness (OR) will be assessed via survey (Readiness for Organizational Change Scale; ROCS). ROCS includes 25 items, each scored on a 5-point scale (1= strongly disagree to 5=strongly agree). Higher mean scores indicate greater organizational readiness for change.
Organizational Readiness (OR) (interview/focus group) | 0, 3-months
  Organizational readiness (OR) will be assessed via interview.

CONTACTS AND LOCATIONS:
Overall Officials: Heather A McKay, PhD, Principal Investigator — University of British Columbia; Joanie Sims Gould, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Centre for Hip Health and Mobility, Robert H.N. Ho Research Centre, University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] Lau, E. Y., Wandersman, A.H., & Pate, R. R. Factors Influencing Implementation of Youth Physical Activity Interventions: An Expert Perspective. Translational Journal of the ACSM: July 1, 2016 - Volume 1 - Issue 7 - p 60-70 doi: 10.1249/TJX.0000000000000006
- [Background] Lubben J, Blozik E, Gillmann G, Iliffe S, von Renteln Kruse W, Beck JC, Stuck AE. Performance of an abbreviated version of the Lubben Social Network Scale among three European community-dwelling older adult populations. Gerontologist. 2006 Aug;46(4):503-13. doi: 10.1093/geront/46.4.503. PMID 16921004
- [Background] Marshall AL, Miller YD, Burton NW, Brown WJ. Measuring total and domain-specific sitting: a study of reliability and validity. Med Sci Sports Exerc. 2010 Jun;42(6):1094-102. doi: 10.1249/MSS.0b013e3181c5ec18. PMID 19997030
- [Background] Rejeski WJ, Rushing J, Guralnik JM, Ip EH, King AC, Manini TM, Marsh AP, McDermott MM, Fielding RA, Newman AB, Tudor-Locke C, Gill TM; LIFE Study Group. The MAT-sf: identifying risk for major mobility disability. J Gerontol A Biol Sci Med Sci. 2015 May;70(5):641-6. doi: 10.1093/gerona/glv003. Epub 2015 Feb 13. PMID 25680917
- [Background] Simonsick EM, Newman AB, Visser M, Goodpaster B, Kritchevsky SB, Rubin S, Nevitt MC, Harris TB; Health, Aging and Body Composition Study. Mobility limitation in self-described well-functioning older adults: importance of endurance walk testing. J Gerontol A Biol Sci Med Sci. 2008 Aug;63(8):841-7. doi: 10.1093/gerona/63.8.841. PMID 18772472
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Veroff, J., Kulka, R. A., & Douvan, E. A. M. (1981). Mental health in America: patterns of help-seeking from, 1957 to 1976: patterns of help-seeking from 1957 to 1976. Basic Books.
- [Background] Warburton, D. E., Jamnik, V. K., Bredin, S. S., & Gledhill, N. (2011). The physical activity readiness questionnaire for everyone (PAR-Q+) and electronic physical activity readiness medical examination (ePARmed-X+). The Health & Fitness Journal of Canada, 4(2), 3-17.
- [Background] Ware, J. E. (1989). SF-36 health status questionnaire. Boston, MA: Institute for the Improvement of Medical Care and Health, New England Medical Center Hospital, Quality Quest Inc.
- [Background] Milton K, Bull FC, Bauman A. Reliability and validity testing of a single-item physical activity measure. Br J Sports Med. 2011 Mar;45(3):203-8. doi: 10.1136/bjsm.2009.068395. Epub 2010 May 19. PMID 20484314
- [Background] Holt, D.T., Armenakis, A.A., Feild, H.S., & Harris, S.G. Readiness for Organizational Change: the systematic development of a scale. The Journal of Applied Behavioral Science. 2007; 43(2): 232-255. https://doi.org/10.1177/0021886306295295
- [Background] Vancouver Coastal Health, Fraser Health, University of British Columbia. My Health My Community Survey. 2014. https://myhealthmycommunity.org/
- [Derived] Nettlefold L, Macdonald HM, Sims Gould J, Bauman A, Szewczyk Z, McKay HA. Does optimizing Choose to Move - a health-promoting program for older adults - enhance scalability, program implementation and effectiveness? Int J Behav Nutr Phys Act. 2024 Dec 18;21(1):140. doi: 10.1186/s12966-024-01649-9. PMID 39695643
- [Derived] Gray SM, Nettlefold L, Mackey D, Gould JS, McKay HA. Feasibility of a Virtual Health-Promoting Intervention (Choose to Move) for Older Adults: A Rapid Adaptation in Response to COVID-19. J Aging Phys Act. 2023 Aug 3;31(6):1003-1015. doi: 10.1123/japa.2023-0011. Print 2023 Dec 1. PMID 37536680